CLINICAL TRIAL: NCT01610466
Title: Design and Validation of a Simulation-based Training Curriculum for Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Royal College of Physicians and Surgeons of Canada (Other)
Responsible Party: Principal Investigator, Teodor Grantcharov, Associate Professor, Department of Surgery, Unity Health Toronto
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: SMH 11-202
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: Education; Simulation; Technical skills training; Laparoscopy; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curriculum training group (Experimental): Surgical residents in the curriculum training group will complete the entire curriculum. They will participate in a cognitive component, which will consist of self-directed readings and a faculty-led seminar. Participants will also train to proficiency in laparoscopic jejunojejunostomy and gastrojejunostomy using a laparoscopic box trainer with cadaveric porcine bowels. Finally, for the non-technical skills component participants will participate in an introductory lecture on non-technical skills in surgery, as well as a practice crisis scenario with a debriefing session.
  Interventions: Procedure: Laparoscopic bariatric surgery ex-vivo training curriculum
- Conventional training group (No Intervention): Participants in the conventional training group will proceed through surgical residency training in the usual fashion.

INTERVENTIONS:
Procedure: Laparoscopic bariatric surgery ex-vivo training curriculum — The training curriculum will consist of a cognitive, technical and non-technical components. Cognitive component will consist of self-directed readings and a faculty-led seminar. Technical component will consist of training to proficiency on cadaveric porcine laparoscopic jejunojejunostomy and gastrojejunostomy models. Non-technical component will consist of an introductory lecture on non-technical skills in surgery and a simulated crisis scenario with a debriefing session.
  Arms: Curriculum training group

SUMMARY:
Laparoscopic bariatric surgery is an advanced laparoscopic procedure with a potential for significant morbidity and mortality along the early part of a surgeon's learning curve. Simulation-based training has been shown to improve a surgeon's technical performance and shorten the learning curves in the operating room. Despite these benefits, there is no evidence-based ex-vivo training curriculum for laparoscopic bariatric surgery. The purpose of this study is to design and validate such a curriculum. This curriculum will include cognitive training, technical laparoscopic skills training (laparoscopic gastrojejunostomy and jejunojejunostomy) and non-technical skills training in a simulated environment. The investigators will assess the effectiveness of the proposed curriculum by conducting a randomized single blinded controlled trial. Cognitive knowledge (multiple choice test), technical skills (performance of a procedure in the operating room) and non-technical skills (performance in a simulated crisis scenario in a simulated environment) will be compared between curriculum trained and conventionally trained groups. The investigators hypothesize that curriculum trained group will have superior knowledge, technical skill and non-technical skills compared to conventionally trained group.

DETAILED DESCRIPTION:
OBJECTIVE: To design and validate a proficiency-based ex-vivo training curriculum for laparoscopic bariatric surgery.

BACKGROUND: Laparoscopic bariatric surgery is an advanced laparoscopic procedure with a potential for significant morbidity and mortality along the early part of a surgeon's learning curve. Simulation-based training has been shown to improve a surgeon's technical performance and shorten the learning curves in the operating room. Despite these benefits, specific simulation-based training curricula have not been widely adopted in residency training programs. This is likely a result of the lack of valid simulation-based training curricula for minimally invasive operations. Presently, there is no evidence-based ex-vivo training curriculum for laparoscopic bariatric surgery. The purpose of this project is to develop and validate such a curriculum.

HYPOTHESIS: Completion of the proposed training curriculum is expected to result in superior cognitive knowledge, superior technical skills in the operating room, and superior performance in a simulated crisis scenario when compared to standard residency training.

METHODS: The evidence-based training curriculum will be made up of cognitive, technical, and non-technical components. The cognitive component will deliver procedure-specific knowledge, while the technical component will provide training in basic and procedure-specific laparoscopic skills. Non-technical component will address additional components of surgical competency including situation awareness, decision making, task management, leadership, communication and teamwork. Technical skills will be learned on a bench-top cadaveric porcine models. Training will follow a distributed practice schedule until preset proficiency benchmarks are achieved. The proposed training curriculum will be validated in a single-blinded randomized controlled trial comparing procedure-specific knowledge, technical performance in the operating room, and non-technical skills in a simulated crisis scenario for 12 surgical residents in the curricular training group and 12 residents in the standard residency training group. Cognitive knowledge will be assessed with a multiple choice examination. Technical performance will be assessed with previously validated procedure-specific and global rating scales. Non-technical skills will be assessed using a previously validated NOTECHS scale.

CONCLUSIONS: The design and implementation of the proposed training curriculum has the potential to affect surgical training programs on a national and international level by standardizing the proficiency of surgical trainees prior to the start of operating room training. This standardization is expected to shorten the learning curves and improve patient safety in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Resident in general surgery at the University of Toronto
* Post - graduate year (PGY) 3 or 4
* Performed less than 10 laparoscopic bariatric operations independently

Exclusion Criteria:

* Residents in other surgical programs at University of Toronto
* Residents in general surgery at the University of Toronto in PGY1, 2, 5 or attending surgeons
* Residents who have performed great than 10 laparoscopic bariatric operations independently

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Difference in operating room performance between curriculum trained and conventionally trained groups | 5 months
  Surgical residents participating in the study will perform a laparoscopic jejunojejunostomy in the operating room. The procedure will be video-recorded through the laparoscopic camera. The videos will be given to a blinded and trained rater who will assess the technical proficiency of the resident using a validated rating scale.

SECONDARY OUTCOMES:
Difference in cognitive knowledge between curriculum trained and conventionally trained groups | 5 months
  Surgical residents in both groups will complete a multiple choice test designed to assess their knowledge in regards to the laparoscopic bariatric surgery.
Difference in non-technical skills between curriculum trained and conventionally trained groups | 5 months
  Surgical residents will participate in a simulated operating room crisis scenario. Their performance will be video recorded and assessed by a trained rater using a validated rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Teodor P Grantcharov, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Zevin B, Aggarwal R, Grantcharov TP. Simulation-based training and learning curves in laparoscopic Roux-en-Y gastric bypass. Br J Surg. 2012 Jul;99(7):887-95. doi: 10.1002/bjs.8748. Epub 2012 Apr 18. PMID 22511220
- [Background] Rehrig ST, Powers K, Jones DB. Integrating simulation in surgery as a teaching tool and credentialing standard. J Gastrointest Surg. 2008 Feb;12(2):222-33. doi: 10.1007/s11605-007-0250-8. Epub 2007 Nov 15. PMID 18004630
- [Background] Aggarwal R, Grantcharov TP, Darzi A. Framework for systematic training and assessment of technical skills. J Am Coll Surg. 2007 Apr;204(4):697-705. doi: 10.1016/j.jamcollsurg.2007.01.016. No abstract available. PMID 17382230
- [Background] Fried GM, Feldman LS, Vassiliou MC, Fraser SA, Stanbridge D, Ghitulescu G, Andrew CG. Proving the value of simulation in laparoscopic surgery. Ann Surg. 2004 Sep;240(3):518-25; discussion 525-8. doi: 10.1097/01.sla.0000136941.46529.56. PMID 15319723
- [Background] Aggarwal R, Boza C, Hance J, Leong J, Lacy A, Darzi A. Skills acquisition for laparoscopic gastric bypass in the training laboratory: an innovative approach. Obes Surg. 2007 Jan;17(1):19-27. doi: 10.1007/s11695-007-9001-x. PMID 17355764
- [Background] Catchpole K, Mishra A, Handa A, McCulloch P. Teamwork and error in the operating room: analysis of skills and roles. Ann Surg. 2008 Apr;247(4):699-706. doi: 10.1097/SLA.0b013e3181642ec8. PMID 18362635
- [Background] Sevdalis N, Davis R, Koutantji M, Undre S, Darzi A, Vincent CA. Reliability of a revised NOTECHS scale for use in surgical teams. Am J Surg. 2008 Aug;196(2):184-90. doi: 10.1016/j.amjsurg.2007.08.070. Epub 2008 Jun 16. PMID 18558392
- [Background] Korndorffer JR Jr, Dunne JB, Sierra R, Stefanidis D, Touchard CL, Scott DJ. Simulator training for laparoscopic suturing using performance goals translates to the operating room. J Am Coll Surg. 2005 Jul;201(1):23-9. doi: 10.1016/j.jamcollsurg.2005.02.021. PMID 15978440